CLINICAL TRIAL: NCT04866784
Title: TENS for Patients With Chronic Testicular Pain (ICO)
Brief Title: TENS for Testicular Pain (ICO): A Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jennifer E. Lee (Other)
Responsible Party: Sponsor-Investigator, Jennifer E. Lee, Adjunct Assistant Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 202004356
Record Dates: First submitted 2020-12-22; First posted 2021-04-30 (Actual); Last update posted 2022-06-23 (Actual); Status verified 2022-06

CONDITIONS: Pain Management
Keywords: Transcutaneous electric nerve stimulation; Idiopathic chronic orchialgia; Testicular Pain; Chronic Pain; Testicular; Scrotum
MeSH Terms: conditions — Agnosia; Chronic Pain | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Intervention Model Description: The study is a prospective, randomized, double-blinded and placebo-controlled crossover design (all participants complete each of the 3 conditions) with randomization to: 1) Active TENS; 2) Placebo TENS; or 3) No Treatment Control. Each subject will receive the 3 TENS treatments in randomized order (one visit per week in three separate weeks). The visits do not have to take place in three consecutive weeks (will depend on participant scheduling preferences), but all three visits must take place within one year
Who Masked: Participant, Outcomes Assessor
Masking Description: The experimenter and subject will be blinded to the treatment conditions. A second experimenter will administer the Active or Placebo TENS, or the Control to ensure appropriate blinding (to ensure no bias from knowing which TENS condition is given at each visit).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- High Sensation TENS (Experimental): Active TENS is delivered for 30mins at a frequency of 100 Hz and pulse duration of 100μsec using the EMPI Select TENS unit (calibrated using an oscilloscope prior to study). The intensity will be increased until patients feel a "maximally strong but comfortable sensation" to ensure an analgesic effect.
  Interventions: Device: Transcutaneous Electrical Nerve Stimulation (TENS)
- Low Sensation TENS (Placebo Comparator): Placebo TENS parameters will be identical to Active TENS (100 Hz and 100 μsec), but a novel placebo TENS unit, previously tested and validated will be used (Rakel et al., 2010). The placebo device provides a current for 30sec and ramps off over 15sec to zero output. An indicator light remains on so it appears to the subject that the unit is still producing current. This unit has demonstrated nearly 100% blinding of investigators such that the investigator applying the TENS is unable to distinguish between the active and the placebo unit; approximately ~50% of subjects are successfully blinded using this unit.
  Interventions: Device: Transcutaneous Electrical Nerve Stimulation (TENS)
- No Treatment Control (No Intervention): The No Treatment Control includes application of TENS electrodes identical to the other 2 conditions, but the unit remains off. This condition will control for potential effects of repeat testing and any placebo effect.

INTERVENTIONS:
Device: Transcutaneous Electrical Nerve Stimulation (TENS) — Transcutaneous electrical nerve stimulation (TENS) is a non-pharmacologic intervention for acute and chronic pain. This treatment involves the application of electric current through the skin; it is safe, easy to use, and inexpensive
  Arms: High Sensation TENS; Low Sensation TENS

SUMMARY:
Idiopathic Chronic Orchialgia (i.e., testicular pain) is a challenging condition to treat, with unresolved testicular pain leading to distress, diminished activities of daily living and decreased quality of life. Testicular Pain may be caused by a tumor, hernia, infection, trauma, vein compression, cysts, and/or postoperative or radiating pain, though is often times unknown. Non-pharmacologic, conservative pain reduction interventions include heat, ice, scrotal support, physical therapy, and/or counseling, and should often be used as first line of defense. More aggressive, invasive, and non-conservative medical treatment options include medications, nerve blocks, and/or surgery, each of which may be effective, but may be invasive and/or cause serious side effects. However, there is no standard of care for managing the testicular pain and many men do not respond to current biomedical or nonpharmacologic treatment options. Novel, non-invasive treatment options are needed for ICO to improve distress, daily living activities, and quality of life. Transcutaneous electrical nerve stimulation (TENS) is a non-pharmacologic intervention for acute and chronic pain. This treatment involves the application of electric current through the skin; it is safe, easy to use, and inexpensive. Despite the impact and distress associated with Testicular Pain, only one known study examined the efficacy of TENS for this condition. A 2018 double-blind, randomized controlled study of people with Testicular Pain reported that TENS improved pain and quality of life significantly more than the control condition (analgesia only). This 2018 study lacked a placebo control condition (i.e., unknown whether pain relief was due to the placebo effect, where knowing an intervention is happening leads to an expectation that pain will decrease, and therefore pain perception decreases independent of the intervention). Thus, the aim of this study is to examine the efficacy of TENS on Testicular Pain using a randomized, placebo-controlled design. The results of this study will be used to inform a larger, federally-funded study.

i. Primary Aim: To assess the efficacy of TENS for Testicular Pain

ii. Secondary Aim: To assess the feasibility of TENS for Testicular Pain

iii. Third Aim: To assess the tolerability of TENS for Testicular Pain

iii. To assess associations between dispositional pain catastrophizing on responsiveness to the TENS intervention.

DETAILED DESCRIPTION:
The overall aim of this study is to examine the efficacy of TENS on Testicular Pain using a randomized, placebo-controlled design. The results of this study will be used to inform a larger, federally-funded study. The study is a prospective, randomized, double-blinded and placebo-controlled crossover design (each participant completes all 3 study conditions) with randomization to 3 study conditions: 1) Active TENS; 2) Placebo TENS; or 3) No Treatment Control. Subjects will be tested 1x/week for 3 weeks. Each subject will receive the 3 treatments in randomized order. Importantly, the experimenter and subject will be blinded to the treatment condition. A second experimenter will administer the Active or Placebo TENS, or the Control to ensure appropriate blinding (to ensure no bias from knowing which TENS condition is given at each visit).

Participants. Thirty men with Testicular Pain (lasting >3 months), aged 18-99yrs will be recruited. Exclusion criteria includes: pain intensity rating ≤ 3/10, contraindications for TENS (pacemaker) or TENS use ≤ 5 years. Participants will provide written informed consent, as approved by the University of Iowa Biomedical Institutional Review Board. TENS Treatment. All subjects will receive each of the 3 TENS treatment conditions while sitting in an upright position. Four adhesive electrodes (2in x 2in) will be placed bilaterally on the: 1) sacrum (for pudendal nerve); and 2) groin (ilioinguinal nerve).

Active TENS includes high frequency TENS delivered for 30mins at a frequency of 100 Hz and pulse duration of 100μsec using the EMPI Select TENS unit (calibrated using an oscilloscope prior to study). The intensity will be increased until patients feel a "maximally strong but comfortable sensation" to ensure an analgesic effect.

Placebo TENS parameters will be identical to Active TENS (100 Hz and 100 μsec), but a novel placebo TENS unit, previously tested and validated will be used. The placebo device provides a current for 30sec and ramps off over 15sec to zero output. An indicator light remains on so it appears to the subject that the unit is still producing current. This unit has demonstrated nearly 100% blinding of investigators such that the investigator applying the TENS is unable to distinguish between the active and the placebo unit; approximately ~50% of subjects are successfully blinded using this unit.

The No Treatment Control includes application of TENS electrodes identical to the other 2 conditions, but the unit remains off. This condition will control for potential effects of repeat testing and any placebo effect.

Patient Measures. Pain will be assessed before and after TENS each session to measure any within visit changes in pain from the TENS intervention. Pain change will be measured using the: 1) Short-Form McGill Pain Questionnaire 27 with qualitative (i.e., sharp, distressing) and quantitative pain scales; and 2) 10-point numeric pain intensity rating scale (NRS) ranging from 0 (no pain) to 10 (worst pain imaginable); These pain measures are valid and reliable. Pain medication intake will also be assessed. Finally, pain-related catastrophizing (i.e., coping) will be measured using the Pain Catastrophizing Scale to determine if any responsiveness to TENS intervention is related to dispositional catastrophizing (i.e., their general catastrophizing levels prior to initiating the TENS study interventions).

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 years to 99;
2. Diagnosis of Idiopathic Chronic Orchialgia (ICO)
3. English Speaking (does not need to be native language)

Exclusion Criteria:

1. Pain intensity rating less than 2/10 at time of first session
2. Inability to read or write
3. Inability to follow directions

4 .Contraindications for TENS (Nickel allergy, pacemaker, open wound in TENS application area)

5. TENS use in last 5 years.

Ages: 18 Years to 99 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Only individuals with at least one descended testicle.
Enrollment: 8 (Actual)
Dates: Start 2020-12-23 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Change in Short-Form McGill Pain Questionnaire (MPQ) Pain Scores | This outcome measure will be used within 10 minutes of the start of each visit (right before TENS is applied) and 30 minutes after TENS is applied (within visit MPQ change) to assess the within visit change in MPQ pain.
  Qualitative (e.g.sharp, distressing) and quantitative pain scales. Quantitative pain scale consists of 15 descriptors (11 sensory, 4 affective) which are rated on an intensity scale of 0 = none, 1=mild, 2=moderate, 3=severe.
Change in 10-point Numeric Pain Intensity Rating Scale (NRS) pain scores | This outcome measure will be used within 10 minutes of the start of each visit (right before TENS is applied) and 30 minutes after TENS is applied (within visit NRS change) to assess the within visit change in NRS pain.
  Quantitative pain scale ranging from 0 (no pain) to 10 (worst pain imaginable)

SECONDARY OUTCOMES:
Pain Catastrophizing Scale (PCS) | This outcome measure will be used at the start of the study (after they consent; baseline). PCS scores range from 0-52 and higher scores mean worse catastrophizing. A decrease in PCS scores is a good outcome.
  Measurement of pain-related coping

CONTACTS AND LOCATIONS:
Overall Officials: Amy M Pearlman, MD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Levine L. Chronic orchialgia: evaluation and discussion of treatment options. Ther Adv Urol. 2010 Oct;2(5-06):209-14. doi: 10.1177/1756287210390409. PMID 21789076
- [Background] Granitsiotis P, Kirk D. Chronic testicular pain: an overview. Eur Urol. 2004 Apr;45(4):430-6. doi: 10.1016/j.eururo.2003.11.004. PMID 15041105
- [Background] Belanger GV, VerLee GT. Diagnosis and Surgical Management of Male Pelvic, Inguinal, and Testicular Pain. Surg Clin North Am. 2016 Jun;96(3):593-613. doi: 10.1016/j.suc.2016.02.014. PMID 27261797
- [Background] Kavoussi PK, Costabile RA. Orchialgia and the chronic pelvic pain syndrome. World J Urol. 2013 Aug;31(4):773-8. doi: 10.1007/s00345-013-1092-5. Epub 2013 May 5. PMID 23645410
- [Background] Masarani M, Cox R. The aetiology, pathophysiology and management of chronic orchialgia. BJU Int. 2003 Mar;91(5):435-7. doi: 10.1046/j.1464-410x.2003.04094.x. No abstract available. PMID 12603394
- [Background] Tojuola B, Layman J, Kartal I, Gudelogul A, Brahmbhatt J, Parekattil S. Chronic orchialgia: Review of treatments old and new. Indian J Urol. 2016 Jan-Mar;32(1):21-6. doi: 10.4103/0970-1591.173110. PMID 26941490
- [Background] Lee JE, Anderson CM, Perkhounkova Y, Sleeuwenhoek BM, Louison RR. Transcutaneous Electrical Nerve Stimulation Reduces Resting Pain in Head and Neck Cancer Patients: A Randomized and Placebo-Controlled Double-Blind Pilot Study. Cancer Nurs. 2019 May/Jun;42(3):218-228. doi: 10.1097/NCC.0000000000000594. PMID 29649082
- [Background] Osiri M, Welch V, Brosseau L, Shea B, McGowan J, Tugwell P, Wells G. Transcutaneous electrical nerve stimulation for knee osteoarthritis. Cochrane Database Syst Rev. 2000;(4):CD002823. doi: 10.1002/14651858.CD002823. PMID 11034768
- [Background] Tantawy SA, Kamel DM, Abdelbasset WK. Does transcutaneous electrical nerve stimulation reduce pain and improve quality of life in patients with idiopathic chronic orchialgia? A randomized controlled trial. J Pain Res. 2017 Dec 27;11:77-82. doi: 10.2147/JPR.S154815. eCollection 2018. PMID 29343983